CLINICAL TRIAL: NCT06014866
Title: ConductIoN System pacInG witH IngeviTy+ for the Left Bundle Branch Area
Brief Title: Conduction System Pacing With INGEVITY+
Acronym: INSIGHT-LBBA
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: Pro00113475
Record Dates: First submitted 2023-08-22; First posted 2023-08-28 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2024-12

CONDITIONS: Bradycardia
Keywords: Conduction system pacing; Cardiac physiologic pacing
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- LBBA INGEVITY+ Pacing: Patients indicated for anti-bradycardia pacing that have been implanted with an INGEVITY+ lead in the LBBA.
  Interventions: Device: Cardiac pacing

INTERVENTIONS:
Device: Cardiac pacing — Patient's previously implanted with the INGEVITY+ lead located in the LBBA

SUMMARY:
The study is intended to evaluate the safety and effectiveness of the Boston Scientific INGEVITY+ cardiac pacing lead when implanted in the left bundle branch area (LBBA).

DETAILED DESCRIPTION:
INSIGHT is a prospectively defined analysis of INGEVITY+ leads that have been previously implanted in the LBBA for the purpose of anti-bradycardia pacing. The results will provide complication free rate (safety) and lead measurements (performance).

Data will be gathered by means of a retrospective, multi-center, US only observational chart review to obtain data on INGEVITY+ leads implanted in the LBBA. Additional data will be gathered from the pulse generator and from the LATITUDE remote monitoring system for pacing thresholds and R-wave amplitude. Consecutive implants will be collected from each site for evaluating the endpoints.

ELIGIBILITY:
Inclusion Criteria for Primary Analysis:

* De novo anti-bradycardia pacing pacemaker implant.
* INGEVITY+ lead implant attempt in the LBBA as documented in the medical record at least 90 days ago.
* LBBAP implant attempt employed a Boston Scientific SSPC series sheath

Exclusion Criteria for Primary Analysis:

-ICD and CRT-D devices

Min Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients implanted with an INGEVITY+ lead implanted in the LBBA to provide rate support for bradycardia.
Sampling Method: Probability Sample
Enrollment: 1383 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2024-08-27 (Actual)

PRIMARY OUTCOMES:
Lead-Related Complication Free Rate | Implant through 90 days
  Adverse events that require correction with an invasive intervention or resulted in significant loss of device functionality.
Pacing Threshold | Implant through 90 days
  Percent of INGEVITY+ leads with pacing capture threshold measurement of less than or equal to 2V.
Sensed R-wave amplitude | Implant through 90 days
  Percent of INGEVITY+ leads with an R-wave amplitude greater than 5mV.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Friedman, MD, Principal Investigator — Duke University
Locations (8):
- United States (8):
  - Sarasota Memorial Health Care System, Sarasota, Florida
  - University of Chicago, Chicago, Illinois
  - Community Heart And Vascular Hospital, Indianapolis, Indiana
  - Essentia Health - Saint Mary's Duluth Clinic, Duluth, Minnesota
  - NewYork-Presbyterian Queens, Flushing, New York
  - Duke University, Durham, North Carolina
  - TriHealth Bethesda North Hospital, Cincinnati, Ohio
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Friedman DJ, Shadrin I, Goldbarg S, Trulock KM, Patel A, Loring Z, Coles SA, Gandhi G, Upadhyay GA, Wold N, Jones PW, Ruble SB, Weinstock J, Latanich CA. Performance of an active fixation stylet-driven lead in left bundle branch area pacing: Results from INSIGHT-LBBA. Heart Rhythm. 2025 Aug;22(8):2047-2054. doi: 10.1016/j.hrthm.2025.01.041. Epub 2025 Feb 4. PMID 39914662